CLINICAL TRIAL: NCT04795011
Title: Additional Manual Lymph Drainage to Standard Postoperative Rehabilitation Protocol in Primary Total Knee Arthroplasty Patients Improves Postoperative Kinesiophobia, Pain and Quality of Life: Preliminary Clinical Results
Brief Title: Outcomes for Manual Lymphatic Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, PhD Student, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SelcukUEC1
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Manual Lymph Drainage; Kinesiophobia; Pain; Quality of Life
MeSH Terms: conditions — Kinesiophobia; Pain | interventions — Exercise; Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Standard rehabilitation protocol will be administered to the control group. In the standard rehabilitation protocol for the first three days after surgery, 3 sets of exercises will be applied as 10 repetitions. The treatment will be initiated for the patients with tolerable coughing and deep breathing exercises. Active dorsi-plantar flexion of the ankle, isometric contraction for the quadriceps, hamstrings and gluteus maximus, for the knee in the supine position on the bed; active heel shift exercises, straight leg raising and standing knee and hip flexion, active hamstring curling, and self-hamstring stretching will be performed. After the exercise, the morning treatment protocol will be completed with a walker at a tolerable distance. The patient will be given assignment in the form of walking and repetition of morning exercises at a tolerable level at least twice during the day.
  Interventions: Other: exercise
- manual lymphatic drainage group (Experimental): manual lymphatic drainage (MLD) will be applied to the second group (MLD group) in addition to the standard rehabilitation protocol
  Interventions: Other: exercise and manual lymphatic drainage

INTERVENTIONS:
Other: exercise and manual lymphatic drainage — MLD will be launched with simple neck application. Hemodynamics of blood and lower extremity motoring will be increased by combining active bilateral shoulder-twisting with breathing after effleurage. Cervical lymph nodes will be stimulated. Back-up treatment will be applied for the abdominal area. Suction power in the ductus thoracicus will be increased with breathing exercises. Ventral drainage will be applied to the lower extremity in accordance with the surgery of the patient.
  Arms: manual lymphatic drainage group
Other: exercise — range of motion and walking exercise
  Arms: control group

SUMMARY:
In this context, the purpose of our study is to investigate the effect of MLD(manual lymphatic drainage) technique applied in addition to the standard postoperative rehabilitation protocol on pain, kinesophobia and quality of life in early periods in patients undergoing primary TKA(total knee arthroplasty) surgery. Our hypothesis is that the addition of the MLD technique to the standard postoperative rehabilitation protocol will improve the early clinical outcomes of patients undergoing primary TKA. In the future perspective, we anticipate that the data obtained as a result of our study will make a significant contribution to the relevant literature on the early and mid-term ameliorative effects of MLD on postoperative pain, kinesiophobia and quality of life, which will be possibly applied in addition to standard postoperative rehabilitation protocols in patients undergoing primary TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 40-85
* were diagnosed with stage IV gonarthrosis
* planned primary total knee arthroplasty (TKA)
* were evaluated before the operation
* whose informed consents

Exclusion Criteria:

* Patients with postoperative pulmonary thromboembolism or treatment-related complications in the past,
* patients with osteoarthritis secondary bone or joint infections,
* patients with morbid obesity,
* patients with presence of hematological disease and malignancy,
* major cardiac pathology,
* venous insufficiency,
* patients taking high-dose anticoagulants
* patients with communication problems

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | 10 minute
  The scale consists of 17 statements. Each statement contains the answers to strongly disagree, disagree, agree, strongly agree. While scoring according to the 4-point Likert scoring system, items 4, 8, 12, and 16 are subjected to reverse scoring. Scoring ranges from 17-68. As the score increases, the painful patient is considered to have an increase in kinesiophobia
Visual Analog Scale (VAS) | 3 minute
  It will be explained to the patients that "0" means "no pain" and "10" means "unbearable pain" on a 10 cm horizontal line. The patients will be asked to mark the pain of activity on the line with the help of a pencil. The values will be calculated with the help of a ruler in centimeters.
Nottingham Health Profile (NHP) | 10 minute
  The questionnaire consists of 38 questions consisting of 6 main topics, namely, energy level, pain, physical mobility, sleep, social isolation, and emotional reactions. The total score for each subtitle is 100, and the total score is obtained by adding the scores obtained from these subtitles. A low score indicates a high quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No